CLINICAL TRIAL: NCT02831361
Title: A Multinational, Multicenter, Randomized, Placebo-controlled, Parallel Group, Double-Blind, Phase 3 Trial to Evaluate the Efficacy and Safety of Gemigliptin 50 mg q.d Compared With Placebo Added to Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Insulin Alone or on Insulin in Combination With Metformin
Brief Title: Trial to Evaluate the Efficacy and Safety of Gemigliptin Compared With Placebo Added on Insulin Alone or on Insulin in Combination With Metformin in Type 2 DM (ZEUS II Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-DPCL016
Record Dates: First submitted 2016-06-23; First posted 2016-07-13 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemigliptin 50mg (Experimental): the subjects should visit a study site at an interval of 6 weeks during the treatment period for 24 weeks in total
  Interventions: Drug: Gemigliptin; Drug: Metformin; Procedure: Diet/exercise questionnaire
- Gemigliptin 50mg placebo (Placebo Comparator): the subjects should visit a study site at an interval of 6 weeks during the treatment period for 24 weeks in total
  Interventions: Drug: Gemigliptin placebo; Drug: Metformin; Procedure: Diet/exercise questionnaire

INTERVENTIONS:
Drug: Gemigliptin
  Arms: Gemigliptin 50mg
Drug: Gemigliptin placebo
  Arms: Gemigliptin 50mg placebo
Drug: Metformin — For patients who have been taking metformin, the patients who had taken at least 1000 mg of metformin daily and continue the same dosage and administration as before participant in the study
Procedure: Diet/exercise questionnaire — doing exercise with about intermediate intensity(50~70%) for ≥150minutes in total over at least 3 times(every other day) weekly should be recommended and regualr diet without greater changes in life style as much as possible during the whole study period.
  the questionnaire regarding diet/exercise will be collected at -week2, week 1 week 7, week 13, week 19, week 25

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of gemigliptin 50 mg orally administered once daily for 24 weeks compared with placebo in patients with type 2 diabetes mellitus who have inadequate glycemic control on insulin alone or on insulin in combination with metformin stably for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus of ≥19 years of age at the time of Visit 1 (Screening)
2. Patients with HbA1c and FPG values measured at central laboratory satisfying the following conditions at the time of Visit 1(Screening)

   * Patients who had not taken OADs other than metformin within 8 weeks prior to Visit 1(Screening) : 7.0% ≤ HbA1c ≤ 11%, FPG < 270mg/dl
   * Patients who had taken OADs other than metformin within 8 weeks prior to Visit 1(Screening) : 6.5% ≤ HbA1c ≤ 10.5%, FPG < 270mg/dl However, re-test can be carried out only once during the visit window, if the central laboratory values don't meet the criteria mentioned above.
3. Patients who had stably received minimum ≥15 U/day and maximum ≤1 U/kg/day of insulin(long-acting, intermediate-acting or pre-mixed) for 8 weeks prior to Visit 1(Screening) ( 'Stably' is defined as the cases in which mean total daily dose of insulin is adjusted to range between ±10% of the dose used on the day of Visit 1(Screening) for 8 weeks prior to Visit 1(Screening).
4. For patients who have been taking metformin, the patients who had taken at least 1000 mg of metformin daily without dose adjustment for 8 weeks prior to Visit 1(Screening)
5. Patients who are applicable to one of the three in the following.

   1. Surgically infertile patients
   2. Postmenopausal female patients of ≥45 years of age for whom ≥2 years elapsed since their last menstruation
   3. Premenopausal fertile female patients or surgically non-infertile male patients who have agreed to use at least 2 kinds of contraceptive measures (certainly including one of the barrier methods) to avoid pregnancy until 14 days after the last dose of the investigational product

      * Barrier methods: Condom, Diaphragm, Cervical cap(Pessary), Spermicide
      * Hormonal methods: Pills, Injection(Depot), Skin patch, Hormonal implant(Implanon), Vaginal ring
      * Intrauterine Devices(IUDs): Cooper IUD(Loop), Hormonal IUD(Mirena)
      * Natural methods: Basic body temperature, Ovulation period, Coitus interruptus, Abstinence
6. Patients who have signed an informed consent themselves after receiving explanation about the objectives, methods, effects, etc. of the clinical study

   For patients who have gone through the washout period, the inclusion criteria below should be checked at Visit 1-1(Screening).
7. Patients whose HbA1c and FPG measured at Visit 1-1(Screening) are 7.0%~11% and <270 mg/dl, respectively
8. Patients whose mean daily dose of insulin checked at Visit 1-1(Screening) ranges between ±10% of the dose checked at Visit 1(Screening)

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus*, gestational diabetes, or secondary diabetes
2. Patients with Body Mass Index(BMI) >40 kg/m2 at the time of Visit 1(Screening)
3. Patients with a history of the following

   * Patients who had experienced severe hypoglycaemia within 24 weeks prior to Visit 1(Screening) or who had experienced hypoglycaemia at least 3 times a week within 8 weeks prior to Visit 1(Screening)†
   * Patients with a history of diabetic ketoacidosis or hyperosmolar non-ketotic coma within 24 weeks prior to Visit 1(Screening) #
   * Patients with a history of myocardial infarction, unstable angina, and coronary artery bypass graft(CABG) within 24 weeks prior to Visit 1(Screening)
   * Patients with NYHA Class III, IV congestive heart failure or arrhythmia requiring treatment at the time of Visit 1(Screening)
   * Patients whose TSH level is out of the normal range and who have thyroidal dysfunction requiring drug therapy at the time of Visit 1(Screening) (However, those who have been taking thyroid hormone at a fixed dose since previous 4 weeks prior to Visit 1[Screening] and whose TSH level is within the normal range can participate in the study.)
   * Patients with severe infection or severe trauma at the time of Visit 1(Screening)
   * Patients who had had a surgical operation within 4 weeks prior to Visit 1(Screening) (excluding minor surgeries without restriction on food and fluid intake) or who are scheduled to have a significant surgery during the study period
   * Patients with pituitary insufficiency or adrenal insufficiency at the time of Visit 1(Screening)
   * Patients with pulmonary embolism, severe pulmonary dysfunction, or who are susceptible to be accompanied by hypoxemia at the time of Visit 1(Screening)
   * Patients on drug therapy due to gastrointestinal disturbance including dehydration, diarrhea, and vomiting at the time of Visit 1(Screening)#
   * Patients who are positive carriers for hepatitis B virus(HBV), hepatitis C virus(HCV), or human immunodeficiency virus(HIV) at the time of Visit 1(Screening) visit
   * Patients with a history of alcoholism or drug addiction within 1 year prior to Visit 1(Screening)
   * Patients with a history of malignant tumors within 5 years prior to Visit 1(Screening). However, patients with basal cell or squamous cell skin cancer, or in situ cervical cancer treated properly can participate in the study.
   * Patients with end-stage renal disease(ESRD) at the time of Visit 1(Screening)
4. Patients with the outcomes of the laboratory tests performed at Visit 1(Screening) applicable to the criteria below

   * Bilirubin >1.5 × upper limit of normal(ULN)
   * AST/ALT >2.5 × ULN
5. Male and female patients on metformin and with serum creatinine level of ≥1.5 mg/dl and ≥1.4 mg/dl, respectively at the time of Visit 1(Screening)
6. Patients with a history of hypersensitivity reactions to the drugs below

   * Gemigliptin or drugs belonging to dipeptidyl-peptidase4(DPP4) inhibitors
   * Metformin or drugs belonging to biguanides
   * Insulin
7. Patients who were administered the drugs below

   * Patients who had been administered anti-obesity drugs within 12 weeks prior to Visit 1(Screening)
   * Patients who had been administered short-acting or rapid-acting insulin before meals within 8 weeks prior to Visit 1(Screening)
   * Patients who had been administered GLP-1 analogues within 8 weeks prior to Visit 1(Screening)
   * Patients who had been administered warfarin, dicoumarin, and digoxin within 4 weeks prior to Visit 1(Screening)
   * Patients who had been being administered glucocorticoids continuously within 2 weeks prior to Visit 1(Screening) or who are required to take glucocorticoids continuously in the future
   * Patients who are being administered any of the strong CYP3A4 inducers (rifampicin[rifampin], dexamethasone, phenytoin, carbamazepine, rifabutin, phenobarbital) at the time of Visit 1(Screening)*
   * Patients who are being administered cimetidine at the time of Visit 1(Screening)
8. Female patients who are pregnant or lactating
9. Patients who have an experience of participation in another clinical study within 12 weeks prior to Visit1(screening)
10. Patients who are otherwise considered to be ineligible for this study on investigators' judgment For patients who have gone through the washout period, the exclusion criteria below should be checked at Visit 1-1(Screening).
11. Patients whose mean daily dose of insulin during the 8-week washout period which has been beyond ±10% of the dose checked at Visit 1(Screening) for ≥ 12 days or for 5 consecutive days

At Visit 1(Screening) or Visit 1-1(Screening), subjects who meet the inclusion/exclusion criteria can enter the 2-week run-in period along with exercise/diet.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
changes from baseline HbA1c at week 25 | baseline (Visit 2) and week 25 (visit 6)

SECONDARY OUTCOMES:
Responder Rate at week 25 | week 25 (visit 6)
  HbA1c <7% , HbA1c <6.5%
Changes of HbA1c at each visit | baseline(visit 2), week 7(visit 3), week 13(visit 4), week 19(visit 5), week 25(visit 6)
  values of parameters at the corresponding visit - values of parameters at visit 2(baseline)
Changes of FPG at each visit | baseline(visit 2), week 7(visit 3), week 13(visit 4), week 19(visit 5), week 25(visit 6)
  values of parameters at the corresponding visit - values of parameters at visit 2(baseline)
Changes of Fasting serum C-peptide at week 25 | baseline (Visit 2) and week 25 (visit 6)
Changes of HOMA-IR at week 25 | baseline (Visit 2) and week 25 (visit 6)
Changes of HOMA-β at week 25 | baseline (Visit 2) and week 25 (visit 6)

OTHER OUTCOMES:
Changes of Total Cholesterol at week 25 | baseline (Visit 2) and week 25 (visit 6)
Changes of cardiovascular disease parameter at week 25 | baseline (Visit 2) and week 25 (visit 6)
  hsCRP
Changes of body weight at each visit | baseline(visit 2), week 7(visit 3), week 13(visit 4), week 19(visit 5), week 25(visit 6)
  values of parameters at the corresponding visit - values of parameters at visit 2(baseline)
Changes of waist circumference at each visit | baseline(visit 2), week 7(visit 3), week 13(visit 4), week 19(visit 5), week 25(visit 6)
  values of parameters at the corresponding visit - values of parameters at visit 2(baseline)
Changes of total daily dose at each visit | visit 2, visit 3, visit 4, visit 5, visit 6
  values of parameters at the corresponding visit - values of parameters at visit 2(baseline)
Changes of LDL-C at week 25 | baseline (Visit 2) and week 25 (visit 6)
Changes of HDL-C at week 25 | baseline (Visit 2) and week 25 (visit 6)
Changes of Triglyceride at week 25 | baseline (Visit 2) and week 25 (visit 6)

IPD SHARING:
Plan to Share IPD: No